CLINICAL TRIAL: NCT01896882
Title: Effects of Dietary Sodium Restriction in Hemodialysis Patients: Randomized Clinical Trial
Brief Title: Dietary Sodium Restriction in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFRGS and HCPA - 120109
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2012-02

CONDITIONS: Hemodialysis Patients
Keywords: Diet, Sodium-Restricted; Food and Nutrition Education; Renal Dialyisis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Nutritional education on sodium restriction diet.
  Interventions: Other: Sodium restriction
- Control (No Intervention): Standard treatment.

INTERVENTIONS:
Other: Sodium restriction
  Arms: Intervention

SUMMARY:
Excess dietary sodium can lead to poor outcomes, such as hypertension, edema and increased risk for cardiovascular diseases. These complications are associated with end stage renal disease (ESRD) progression and mortality in renal patients. This study aims to evaluate the effects of nutritional counseling restricting dietary sodium and its relation to clinical and diet factors, nutritional knowledge and quality of life in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stable patients on dialysis for at least 3 months, over 18 years old, of both sexes, who agree to participate in the study.

Exclusion Criteria:

* Patients with low cognitive ability, psychiatric disorders, with acute or infectious disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Sodium intake | Baseline, 30, 90, 180 and 360 days
  Sodium intake will be evaluated by food record and a food frequency questionnaire.
Quality of life | Baseline, 180 and 360 days.
  Quality of life will be evaluated by the Brazilian Portuguese version of the Kidney Disease and Quality-of-Life Short-Form (KDQOL-SF) questionnaire.

SECONDARY OUTCOMES:
Interdialytic weight gain | Baseline, 30, 90, 180 and 360 days.
  Will be considered the amount of weight gain between 2 dialysis sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Corrêa Souza, Professor, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil